CLINICAL TRIAL: NCT06746207
Title: Evaluating Patient and Caregiver Satisfaction on the Informed Consent Process in Surgical Practice in a Tertiary Care Centre: a Cross-Sectional Study
Brief Title: Evaluating Patient and Caregiver Satisfaction with the Informed Consent Process in Surgery
Status: Completed | Type: Observational
Sponsor: Maharajgunj Medical Campus (Other)
Responsible Party: Principal Investigator, Asim Shrestha, Principal Investigator, Maharajgunj Medical Campus
Other Study IDs: 225-6-12
Record Dates: First submitted 2024-12-11; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Informed Consent; Patient and Caregiver Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients and Caregivers: This cohort includes two groups: patients undergoing major elective surgery and their caregivers. The patients are asked to provide feedback on their understanding and satisfaction with the informed consent process. The caregivers, who often provide the informed consent on behalf of the patients, are also surveyed to assess their perspectives on the consent process. There is no intervention in this study; the focus is on evaluating perceptions, satisfaction, and the communication process surrounding informed consent in a surgical setting.
  Interventions: Other: Informed Consent Process Evaluation

INTERVENTIONS:
Other: Informed Consent Process Evaluation — This study does not involve a clinical intervention. Instead, it focuses on evaluating the existing process of informed consent in a surgical setting. Patients and caregivers will be surveyed to assess their understanding, satisfaction, and perceptions of the informed consent process. The study examines factors such as clarity of information provided, patient and caregiver involvement, and overall satisfaction with the process, without altering the current practices. The goal is to identify areas for improvement in communication and documentation, ensuring that patient rights and autonomy are respected.

SUMMARY:
The goal of this observational study is to evaluate patient and caregiver satisfaction with the informed consent process in surgical practice at a tertiary care center in Nepal. The main questions it aims to answer are:

How satisfied are patients and caregivers with the current informed consent process in surgery? How well do patients and caregivers understand the informed consent information provided? Are there differences in satisfaction and understanding based on factors such as education level or family involvement? Researchers will compare the perceptions of patients and caregivers to understand if there are gaps in communication and satisfaction.

Participants will:

Complete a structured questionnaire assessing their understanding and satisfaction with the informed consent process.

Share their views on the type and quality of information provided during the consent process.

Rate their satisfaction on a 10-point scale based on their experience with the informed consent procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older undergoing major elective surgical procedures requiring regional or general anesthesia.
* Caregivers of eligible patients who provide informed consent on behalf of the patient.
* Willingness to participate and provide consent for the study.

Exclusion Criteria:

* Patients undergoing emergency surgeries.
* Patients who are unable to participate due to language barriers or cognitive impairment.
* Patients or caregivers who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients undergoing major elective surgeries across various departments, including General Surgery, Neurosurgery, Plastic Surgery, Urology, ENT, Orthopedics, and Obstetrics & Gynecology. Caregivers of these patients, typically responsible for providing informed consent, will also be included. The study aims to capture the perspectives of both groups regarding the informed consent process.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Patient and Caregiver Satisfaction with the Informed Consent Process | Within 24 hours of the surgery
  Satisfaction with the informed consent process will be evaluated using a structured questionnaire. Patients and caregivers will rate satisfaction on a 10-point Likert scale (1 = least satisfied, 10 = most satisfied) and respond to Yes/No questions assessing their understanding of the surgery's nature, risks, long-term effects, and anesthesia-related complications. Additional questions evaluate the clarity and completeness of the consent form, including whether essential components (e.g., patient name, diagnosis, procedure details, and risks) were documented. Responses aim to identify gaps in the consent process and assess whether it meets patient and caregiver expectations, as well as legal and ethical standards.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Medicine, Maharajgunj, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
Since this is an observational study focused on evaluating the informed consent process, Individual Participant Data (IPD) will not be shared as part of the study's results. However, the aggregated findings, such as overall satisfaction scores and analysis of demographic factors influencing consent understanding, will be presented in the final study report.